CLINICAL TRIAL: NCT04598945
Title: Acquisition and Retention of Motor Memories in Adults and Typically Developing Children. IRM f Study
Brief Title: Acquisition and Retention of Motor Memories in Adults and Typically Developing Children
Acronym: MOTORMEMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: TIMC-IMAG (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC20.005
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Memory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adults (Experimental): The subject will be subjected to 2 functional MRI sessions spaced 3 days apart Each session will be composed of the same MRI sequences without injection, namely an anatomical exploration sequence followed by sequences of functional exploration of rest and activation (while the subject performs the task motor). The resting functional exploration sequences will frame (1 before, 1 after) the functional activation sequence.
  Interventions: Other: Functionel MRI
- Children (Experimental): The subject will be subjected to 2 functional MRI sessions spaced 3 days apart Each session will be composed of the same MRI sequences without injection, namely an anatomical exploration sequence followed by sequences of functional exploration of rest and activation (while the subject performs the task motor). The resting functional exploration sequences will frame (1 before, 1 after) the functional activation sequence.
  Interventions: Other: Functionel MRI

INTERVENTIONS:
Other: Functionel MRI — During the activation fMRI sequences, the subject will perform target pointing tasks, that is to say that he will have to reach, by controlling a cursor using a non-magnetic joystick, targets projected onto a display screen. In each of the pointing tasks he will have to reach the target as quickly and as precisely as possible, and stay in the center of it for a long time times reached.

SUMMARY:
Our motor skills require motor memories without which our behavior is only reflexes and stereotypies. The way which these memories form in the human brain constitute therefore a major challenge for neuroscience research. Some a lot of evidence suggests that any new motor skills is acquired in the cerebellum and then persisted in the cortex. This vision seems however caricature, the formation of memories motor probably requiring complex remodeling of cortico-cerebellar networks. The MotorMemo project aspires to better understand this remodeling, by testing more specifically the hypothesis of cerebellar weakening and strengthening cortical as a substrate for the formation of motor memories. A longitudinal study using a sensorimotor adaptation protocol, fMRI as well as a developmental perspective is proposed to verify this hypothesis.

DETAILED DESCRIPTION:
A fundamental human faculty is that of adapting our motor behavior to changing environmental conditions. This faculty is comparable to an apprenticeship adaptive during which the individual updates, on a trial and error basis, the correspondence between sensory inputs and the resulting motor commands. Once updated, these correspondences or internal models allow the individual to produce a behavior precise and reproducible motor. The issue of model acquisition and retention internal movement is therefore central to our understanding of motor control. Relatedly, this question constitutes a gateway to a more comprehensive understanding of the mechanisms of learning and procedural memory.

The MotorMemo project therefore aims to study the formation of internal models of movement in the human brain, with the particularity of being interested in the correlates cerebral processes of acquiring and retaining an internal model of visuomotor transformation in healthy children (8-12 years) and adults.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* affiliated to a social security scheme
* who gave their consent to participate in the study

Exclusion Criteria:

* Contraindication to MRI
* visual impairment;
* suffering from one of the following pathologies:

  * dysphasia,
  * ADHD,
  * dyspraxia,
  * dyslexia,
  * dysorthography,
  * dyscalculia;
  * history of epilepsy
* subject in period of exclusion from another study,
* subject under administrative or judicial supervision
* pregnant or breastfeeding women
* Persons referred to in articles l1121-8

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate, in adults and children, whether the acquisition and retention of a new internal movement pattern are linked to the activation of a large cortico-cerebellar network ladder. | 3 days
  Change in cerebellar activation and cortical induced by the visuomotor adaptation task compared to a task motor control not requiring adaptation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France